CLINICAL TRIAL: NCT01990092
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety and Nutritional Benefits of Metanx® in Subjects With Diabetic Peripheral Neuropathy
Brief Title: The Nutritional Benefits of Metanx in Patients With Diabetic Peripheral Neuropathy (MEDIAN)
Acronym: MEDIAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pamlab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: M-003
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Peripheral Neuropathy; B Vitamin Deficiency
Keywords: Metanx; B vitamins; neuropathy; nutrition
MeSH Terms: conditions — Vitamin B Deficiency | interventions — metanx

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metanx (Experimental): Subjects will take 2 Metanx tablets once daily for 48 weeks.
  Interventions: Other: Metanx
- Placebo (Placebo Comparator): Subjects will take 2 placebo tablets once daily for 48 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Metanx — Metanx is a prescription medical food.
  Arms: Metanx
Other: Placebo
  Arms: Placebo

SUMMARY:
The objectives of the MEDIAN study are to evaluate the short-term and long-term safety and nutritional benefits of Metanx® versus placebo in subjects with mild to moderate diabetic peripheral neuropathy (DPN). Short-term effects will be evaluated during the first 16 weeks of treatment, and long-term effects will be evaluated over the duration of a 48 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female between 25 and 80 years of age, inclusive, at the time of consent
* Have a diagnosis of diabetes mellitus Type 2 as defined by the American Diabetes Association and on stable therapy as defined per the investigator's opinion for at least 1 month before the Screening Visit.
* Have a diagnosis of DPN established at least 6 months but not greater than 7 years prior to Screening
* If receiving DPN-related medication, doses must be stable for at least 6 weeks and should be taking only one of the following medications compliant with Exclusion Criterion 7:

  * Alpha-2-delta ligand [e.g., pregabalin (Lyrica) or gabapentin (Neurontin)
  * Anticonvulsant [e.g., carbamazepine, topiramate (Topamax), valproic acid (Depakote) or lamotrigine (Lamictal)]
  * Serotonin-norepinephrine Reuptake Inhibitor (SNRI) [e.g., duloxetine (Cymbalta) or venlafaxine (Effexor)]
  * Tricyclic antidepressant (TCA) [e.g., amitriptyline, nortriptyline, imipramine, and desipramine (Norpramin, Pertofrane)]
* Have a score between 3 and 6, inclusive, on the Michigan Neuropathy Screening Instrument (MNSI) Part b
* Have a minimum score of 6 on the NTSS-6 at Screening
* Have negative urinalysis for drugs of abuse, such as amphetamines, barbiturates, cannabinoids, cocaine, or opiates
* Have a negative urine pregnancy test at Screening if female and of childbearing potential
* If female, must be either of nonchildbearing potential (surgically sterile or 2 years postmenopausal) or agree to use two methods of effective contraception such as hormonal contraception, intrauterine device or other mechanical contraception device, or condom plus spermicide during the subject's participation
* If male, must be surgically sterile or agree to use two methods of effective contraception such as condom plus spermicide during the subject's participation
* Have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an institutional review board (IRB), and agree to abide by the study restrictions and return to the site for the required assessments
* Have provided written authorization for use and disclosure of protected health information

Exclusion Criteria:

* Be pregnant or lactating
* Have a history of amputation, skin ulceration, and/or active Charcot of either foot
* Have a history of previous surgery involving the spine or lower extremity, with residual symptoms of pain or difficulty with movement
* Have Crohn's disease or a history of any type of bariatric surgery or any surgical resection of all or part of the stomach, duodenum, jejunum, and/or ileum. (Previous surgical resections of the colon that spared the stomach, duodenum, jejunum and ileum are allowed.)
* Have a history of surgery or hospitalization within 2 months prior to Screening or planned hospitalization at any time during the study
* Be taking systemic corticosteroids within 2 months prior to Screening, opiates or tramadol hydrochloride within 6 weeks prior to Screening, and/or immunosuppressives, or receiving radiotherapy within 6 months prior to Screening
* Be taking more than one anticonvulsant, serotonin-norepinephrine reuptake inhibitor (SNRI), or tricyclic antidepressant (TCA)
* Have ongoing evidence of peripheral vascular disease, including greater than one nonpalpable pulse on either foot, history of claudication, or history of lower extremity vascular bypass surgery or angioplasty
* Have circulating glycated hemoglobin (HbA1c) exceeding 11% at Screening
* Have an estimated glomerular filtration rate (eGFR) less than or equal to 40 ml/min using the Modification of Diet in Renal Disease (MDRD) formula at Screening or have end-stage renal disorder requiring hemodialysis
* Have uncontrolled hypertension defined as sustained systolic blood pressure (SBP) greater than 200 mmHg or diastolic blood pressure (DBP) greater than 110 mmHg at screening
* Have lung disease (uncontrolled asthma or shortness of breath) within 2 months prior to Screening
* Use of any of the following supplements within 6 weeks before Screening: evening primrose oil, vitamin B12 injection, greater than 10 mg of vitamin B6, or greater than 800 µg of folate
* Have previously failed two or more prior therapies for painful DPN
* Currently abusing alcohol or drugs or have a history of such abuse within the past 3 years. (Alcohol abuse is defined as more than 2 drink units per day for women and more than 3 drink units per day for men. One drink unit is defined as 1.5 oz [45 mL] of distilled spirits, 5 oz [150 mL] of wine, or 12 oz [360 mL] of beer.)
* Have any nondiabetic cause of peripheral neuropathy
* Have a history of documented lumbar nerve entrapment or symptoms suggestive of a lumbar nerve entrapment
* Have a history of systemic lupus erythematosis, rheumatoid arthritis, Sjögren's syndrome, or mixed connective tissue disease
* If receiving thyroid replacement therapy, should be on a stable dose for at least 6 weeks prior to Screening
* Have a history of a positive HIV test or active Hepatitis B or C infection.
* Have a history or presence of malignancy within 10 years prior to Screening except for basal or squamous cell carcinoma of the skin. Records to be submitted to Pamlab for review and approval to randomize.
* Have prior use of or intolerance to Metanx® or any of its active ingredients
* Have been dosed or used a medical device in another investigational trial within 60 days prior to Screening.
* Have any clinically significant existing medical, psychiatric, or nonmedical condition that in the opinion of the investigator places the subject at undue risk, prevents compliance with the study protocol, or potentially jeopardizes the quality of the data to be generated

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in plasma methylmalonic acid (MMA) levels | 16 weeks

SECONDARY OUTCOMES:
Change in plasma 5-methyltetrahydrofolate levels | 16 weeks
Change in plasma vitamin B6 levels | 16 weeks
Change in plasma vitamin B12 levels | 16 weeks
Change in urine microalbumin/creatinine ratio | 48 weeks
Change in epidermal nerve fiber density | 48 weeks
  This neuropathy-specific measure will be evaluated to monitor for signs of disease progression.
Change in neuropathic disability as measured by the Michigan Neuropathy Screening Instrument part B | 48 weeks
  This neuropathy-specific measure will be evaluated to monitor for signs of disease progression.
Change in neuropathic symptoms as measured by the Neuropathy Total Symptom Score-6questionnaire(NTSS-6) | 16 weeks
  This neuropathy-specific measure will be evaluated to monitor for signs of disease progression.
Change in neuropathic symptoms as measured by the Neuropathy Total Symptom Score-6 questionnaire (NTSS-6) | 48 weeks
  This neuropathy-specific measure will be evaluated to monitor for signs of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (25):
- United States (25):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Meridien Research, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - Florida Medical Clinic, Wesley Chapel, Florida
  - North Chattahoochee Family Physicians, LLC, Johns Creek, Georgia
  - Willis-Knighton Physician Network / WKB Family Medicine Associates, Bossier City, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Urgent Care Specialists, LLC dba Hometown Urgent Care & Occupational Health, Dayton, Ohio
  - CRI Lifetree, Philadelphia, Pennsylvania
  - Trinity Clinical Research, LLC, Tullahoma, Tennessee
  - FutureSearch Trials of Neurology, L.P., Austin, Texas
  - Centex Studies Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Northeast Clinical Research of San Anotnio, LLC, Schertz, Texas
  - ClinPoint Trials, LLC, Waxahachie, Texas
  - Strelitz Diabetes Center, Norfolk, Virginia